CLINICAL TRIAL: NCT04718909
Title: Regorafenib Combined With Sintilimab Versus Regorafenib Alone as the Second-line Treatment for Unresectable Hepatocellular Carcinoma
Brief Title: Regorafenib Plus Sintilimab vs. Regorafenib as the Second-line Treatment for HCC
Acronym: REGSIN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: ZhuHai Hospital (Other); Shenzhen People's Hospital (Other); Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Second Affiliated Hospital of Nanchang University (Other); The First People's Hospital of Zhaoqing (Unknown); Fifth Affiliated Hospital, Sun Yat-Sen University (Other); Cancer Hospital of Guangxi Medical University (Other); Jiangmen Central Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Peking University Shenzhen Hospital (Other); Jieyang People's Hospital (Other); Shantou Central Hospital (Other); Yuebei People's Hospital (Other); Zhaoqing Gaoyao People's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIIR-05
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Hepatocellular Carcinoma Non-resectable
Keywords: Hepatocellular carcinoma; Regorafenib; Sintilimab; Second-line treatment
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — regorafenib; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regorafenib + sintilimab (Experimental): Regorafenib combined with sintilimab.
  Interventions: Drug: Regorafenib + sintilimab
- Regorafenib (Active Comparator): Regorafenib alone.
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib + sintilimab — Regorafenib: 160 mg p.o. qd for 3 weeks of every 4 week cycle (i.e. 3 weeks on, 1 week off).
  Sintilimab: 200mg i.v. q3w.
  Arms: Regorafenib + sintilimab
Drug: Regorafenib — 160 mg p.o. qd for 3 weeks of every 4 week cycle.
  Arms: Regorafenib

SUMMARY:
This study is conducted to evaluate the efficacy and safety of regorafenib plus sintilimab compared with regorafenib alone as the second-line treatment for patients with unresectable hepatocellullar carcinoma (HCC).

DETAILED DESCRIPTION:
This is an open-label, multicenter, randomized controlled trial to evaluate the efficacy and safety of regorafenib plus sintilimab compared with regorafenib alone as the second-line treatment for unresectable HCC.

180 patients with unresectable HCC who progress after sorafenib or lenvatinib treatment or are intolerant to these drugs will be enrolled in the study. The Patients will be treated with regorafenib plus sintilimab or regorafenib alone using an 1:1 randomization scheme.

Regorafenib will last until disease progresses, intolerable toxicity, withdrawal of informed consent, loss of follow-up, death, or other circumstances that require termination of treatment, whichever occurs first. The administration of regorafenib will be delayed in cases of severe toxicities. And after recovery, regorafenib will be reintroduced at a reduced dose according to the dose delay and reduction guidelines. Treatment of sintilimab will last up to 24 months, or until disease progresses, intolerable toxicity, withdrawal of informed consent, loss of follow-up, death, or other circumstances that require termination of treatment, whichever occurs first. In the arm of regorafenib plus sintilimab, patients will be allowed to have regorafenib or sintilimab as a sigle agent and will be still considered on study when the other drug cause intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable HCC confirmed by histology/cytology or clinically.
* Failure to prior sorafenib or lenvatinib treatment, or intolerance to sorafenib or lenvatinib.
* For patients who cannot tolerant to sorafenib or lenvatinib, the AEs must resolve to ≤ grade 1 (NCI-CTCAE v5.0) before randomization.
* Child-Pugh class A.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at enrollment.
* At least one measurable lesion.
* Adequate organ and hematologic function.
* Life expectancy of at least 3 months.
* For women of childbearing potential and for men: agreement to remain abstinent.

Exclusion Criteria:

* Diagnosis of fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC.
* Diffuse HCC.
* Portal vein tumor thrombus (PVTT) involves the main trunk and contralateral branch or upper mesenteric vein.
* Inferior vena cava tumor thrombus.
* Metastatic disease that involves major airways or blood vessels.
* Symptomatic, untreated or progressing central nervous system metastasis.
* History of hepatic encephalopathy
* History of organ and stem cell transplantation
* Uncontrolled ascites, hydrothorax or pericardial effusion
* Patients who receive systemic therapy except for sorafenib and lenvatinib within 4 weeks before randomization, including other molecular targeted drugs, chemotherapy (including hepatic arterial infusion chemotherapy), immunotherapy, and herbal therapy or traditional Chinese medicine with anti-cancer activity.
* Prior esophageal and/or gastric varices bleeding within 6 months prior to initiation of study treatment.
* Untreated or incompletely treated esophageal and/or gastric varices with high-risk for bleeding.
* History of venous thromboembolism, but implantable i.v. ports, catheter-derived thrombosis, superficial venous thrombosis, or thrombosis effectively treated by regular anticoagulant therapy are excluded.
* Use of anticoagulants which need monitoring of international normalized ratio.
* Patients unable to swallow oral medications; Gastrointestinal malabsorption, gastrointestinal anastomosis, or any other condition that may affect the absorption of regorafenib.
* Serious, non-healing or dehiscing wound, active ulcer, or untreated bone fracture underwent major surgery (craniotomy, thoracotomy or open surgery) within 4 weeks; non-recovery from side effects of these procedure.
* Active tuberculosis.
* History of malignancy other than HCC within 5 years prior to screening. Patients with skin basal cell carcinoma, skin squamous cell carcinoma, or carcinoma in situ (e.g., breast carcinoma and cervical carcinoma in situ) who have received potentially curative treatment is allowed.
* Hepatitis B is allowed if no active replication is present. Hepatitis C is allowed if no antiviral treatment is required.
* Co-infection of hepatitis B virus (HBV) and hepatitis C virus (HCV) or HBV and hepatitis D virus (HDV).
* Active infection requiring systemic treatment. Hepatitis B without active replication is allowed. Hepatitis C not requiring antiviral treatment is allowed.
* Use of antibiotics within 2 weeks prior to injection of sintilimab.
* Use of immunosuppressive drugs in the past 4 weeks, excluding the routes of topical glucocorticoids or physiological doses of systemic glucocorticoids (ie no more than 10 mg/day of prednisone or equivalent). Temporary use of glucocorticoids for dyspnea symptoms such as asthma and chronic obstructive pulmonary disease is allowed.
* History of idiopathic pulmonary fibrosis, interstitial pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis.
* Autoimmune disease or immune deficiency.
* Inadequately controlled hypertension; history of hypertensive crisis or hypertensive encephalopathy.
* Female patients who are pregnancy or breastfeeding.
* Other acute or chronic diseases, mental illness, or abnormal laboratory test results that may lead to the following outcomes: increase the risk of participating in study or study drug administration, or interfere with the interpretation of the study results and considered by investigator as "NOT" eligible to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2021-01-09 (Actual); Primary Completion 2023-07-08 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) assessed by investigators according to Response Evalutaion Criteria in Solid Tumors (RECIST) v1.1 and immune-related RECIST (irRECIST) | 24 months
  The time from date of randomization until the first occurrence of disease progression or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Adverse Events (AEs) | 24 months
  Number of patients with AE, treatment-related AE (TRAE), immune-related AE (irAE), AE of special interest (AESI), serious adverse event (SAE), assessed by NCI CTCAE v5.0.
Overall survival (OS) | 24 months
  The time from date of randomization to death due to any cause.
Time to Progression (TTP) assessed by investigators according to RECIST 1.1 and irRECIST | 24 months
  The time from date of randomization until the first occurrence of disease progression.
Objective response rate (ORR) assessed by investigators according to RECIST 1.1 and irRECIST. | 24 months
  The percentage of patients who had a best overall tumor response rating of complete response (CR) or partial response (PR).
Disease control rate (DCR) assessed by investigators according to RECIST 1.1 and irRECIST | 24 months
  The percentage of patients who had a tumor response rating of CR, PR, or stable disease (SD).
PFS assessed by investigators according to Modified RECIST (mRECIST) | 24 months
  The time from date of randomization until the first occurrence of disease progression or death due to any cause, whichever occurs first.
TTP assessed by investigators according to mRECIST. | 24 months
  The time from date of randomization until the first occurrence of disease progression.
ORR assessed by investigators according to mRECIST | 24 months
  The percentage of patients who had a best overall tumor response rating of CR or PR.
DCR assessed by investigators according to mRECIST. | 24 months
  The percentage of patients who had a tumor response rating of CR, PR, or SD.

CONTACTS AND LOCATIONS:
Overall Officials: Kangshun Zhu, Dr., Study Chair — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- the Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China